CLINICAL TRIAL: NCT05530369
Title: The Link Between "Time In Range" Versus HbA1c and the Presence of Chronic COmplications in Type 1 Diabetes: a Longitudinal Study - The TIRCO Study
Brief Title: The Link Between "Time In Range" Versus HbA1c and the Presence of Chronic COmplications in Type 1 Diabetes: a Longitudinal Study
Acronym: TIRCO
Status: Completed | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Sponsor
Other Study IDs: TIRCO
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-08

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Type 1 Diabetes; HbA1c; Time In Range; Chronic complications; Continuous Glucose Monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
HbA1c is currently the only metric of glucose control showing an association with chronic complications of type 1 diabetes mellitus (T1D). Time in range (TIR, 70-180 mg/dL) measured by real-time continuous glucose monitoring (CGM) might be a better marker. In this study, the investigators studied the clinical significance of a 10% increase of TIR over two years.

DETAILED DESCRIPTION:
Adult subjects (age ≥ 18 years) with T1D were consecutively recruited in three multicenter studies (RESCUE, FUTURE, ALERTT1 studies) organized between September 2014 and 19 November 2021. For the TIRCO study, only the data from patients recruited at the University Hospital of Antwerp were analyzed. Initially, the data from 498 patients were collected. Pregnant patients and patients with beta-cell transplantation were excluded from the study, resulting in the inclusion of 479 patients. Consecutive patients starting CGM were proposed to participate and were included into the study after signing informed consent.

The study population consisted of 445 patients who used Freestyle libre, 21 patients who used CGM in hybrid closed loop and 13 patients who used Dexcom G4 and G6, resulting in a total of 479 patients.

In this project, the investigators looked into the link between TIR versus HbA1c and the presence of chronic complications in adults with T1D.

The primary endpoint was to evaluate the link between TIR and the presence of chronic microvascular complications as formulated by the following research question: "What is the clinical significance of a 10% increase of TIR over two years?"

The secondary endpoint was to assess the link between TIR and independent risk factors for micro- and macrovascular complications such as sex, age, BMI, lipids, blood pressure, HbA1c, time in range, mean glucose, diabetes duration, method of insulin administration (MDI or CSII), type of sensor and sensor compliance.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus
* Using Real-Time Continuous Glucose Monitoring (rtCGM), Intermittently Scanned CGM (isCGM) or (Hybrid) Closed Loop (HCL) as diabetes treatment
* Willing to sign informed consent

Exclusion Criteria:

* Pregnancy
* Patients that had beta-cell transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects (age ≥ 18 years) with T1D were consecutively recruited in three multicenter studies (RESCUE, FUTURE, ALERTT1 studies) organized between September 2014 and 19 November 2021. For the TIRCO study, only the data from patients recruited at the University Hospital of Antwerp were analyzed. Initially, the data from 498 patients were collected. Pregnant patients and patients with beta-cell transplantation were excluded from the study, resulting in the inclusion of 479 patients. Consecutive patients starting CGM were proposed to participate and were included into the study after signing informed consent.
  The study population consisted of 445 patients who used Freestyle libre, 21 patients who used Standalone CGM and 13 patients who used Dexcom G4 and G6, resulting in a total of 479 patients.
Sampling Method: Probability Sample
Enrollment: 479 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Time In Range (TIR, 70-180 mg/dL) | 12 months
  Change in time spent in range (70-180 mg/dL) from baseline to 12 months
Time In Range (TIR, 70-180 mg/dL) | 24 months
  Change in time spent in range (70-180 mg/dL) from baseline to 24 months; Change of 10% in time spent in range (70-180 mg/dL) compared from baseline to 24 months
Diabetic eye disease | 12 months
  Change in presence of microvascular complication 'Diabetic eye disease' (preproliferative retinopathy, proliferative retinopathy, maculopathy) from baseline to 12 months
Diabetic eye disease | 24 months
  Change in presence of microvascular complication 'Diabetic eye disease' (preproliferative retinopathy, proliferative retinopathy, maculopathy) from baseline to 24 months
Nephropathy | 12 months
  Change in presence of microvascular complication 'Nephropathy' (albuminuria
  ≥ 20µg/min or eGFR < 60 ml/min/1,73m^2) from baseline to 12 months
Nephropathy | 24 months
  Change in presence of microvascular complication 'Nephropathy' (albuminuria
  ≥ 20µg/min or eGFR < 60 ml/min/1,73m^2) from baseline to 24 months
Neuropathy | 12 months
  Change in presence of microvascular complication 'Neuropathy' (monofilament score < 12/12) from baseline to 12 months
Neuropathy | 24 months
  Change in presence of microvascular complication 'Neuropathy' (monofilament score < 12/12) from baseline to 24 months

SECONDARY OUTCOMES:
HbA1c (%) | 12 months
  Change in HbA1c from baseline to 12 months
HbA1c (%) | 24 months
  Change in HbA1c from baseline to 24 months
Mean glucose (mg/dl) | 12 months
  Change in mean glucose (mg/dl) from baseline to 12 months
Mean glucose (mg/dl) | 24 months
  Change in mean glucose (mg/dl) from baseline to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Christophe De Block, MD, PhD, Principal Investigator — University Hospital, Antwerp

IPD SHARING:
Plan to Share IPD: No